CLINICAL TRIAL: NCT00189579
Title: A Phase II Study Designed to Evaluate the Safety and Efficacy of the Addition of Herceptin to a Carboplatin-Paclitaxel Regimen in Early Relapse Patients (< 6 Months) With Ovarian Cancer, Overexpressing HER2, Previously Treated With Carboplatin-Paclitaxel
Brief Title: Addition of Herceptin to a Carboplatin-Paclitaxel Regimen in Patients With Ovarian Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCHERCEPTIN1
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-08-17 (Estimated); Status verified 2007-08

CONDITIONS: Ovarian Cancer
Keywords: HERCEPTIN; Carboplatin; Paclitaxel; Relapse
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — Trastuzumab

INTERVENTIONS:
Drug: Herceptin

SUMMARY:
The purpose of this study is to evaluate whether or not the addition of Herceptin may be of benefit to a standard regimen of carboplatin-paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older; patients with histologically proven diagnosis of ovarian cancer.
* Patients with metastatic disease and an overexpression of HER2 (as determined by immunochemistry)
* Patients who have progressed while receiving treatment, or within 6 months after completion of treatment. Patients must have received carboplatin and paclitaxel.
* Patients who have received at minimum one line of chemotherapy
* 3 weeks minimum since last treatment with chemotherapy must have elapsed
* Patients must have at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) or an assessable cancer antigen (CA) 125 > 1.25 x upper limit of normal (ULN)
* Patients must have ECOG of 2 or less
* Left ventricular ejection fraction (LVEF) of 50% or better
* Patients have given their signed and verbal consent

Exclusion Criteria:

* Previous treatment with Herceptin or similar products affected growth factors (eg: Iressa)
* Another experimental treatment in the previous 30 days
* No overexpression of HER2 receptors
* Patients having received high-dose chemotherapy or stem-cell interventions
* Other cancers within the last 5 years
* Patients with dyspnea at rest or requiring oxygen therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Pujade-Lauraine, MD, PhD, Study Chair — Hopital Hotel-Dieu
Locations (1):
- Hopital Hotel-Dieu, Paris, France